CLINICAL TRIAL: NCT05097846
Title: Comparison of Vonoprazan Fumarate-based Triple Therapy Versus Proton Pump Inhibitor and Bismuth Based Quadruple Therapy in the Eradication of Helicobacter Pylori: a Single-center Prospective Open-label Controlled Study
Brief Title: Differences in the Eradication of Helicobacter Pylori by Different Therapies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: wang xiaoyan (Other)
Responsible Party: Sponsor-Investigator, wang xiaoyan, Director, Head of Gastroenterology, Principal Investigator, Clinical Professor, The Third Xiangya Hospital of Central South University
Organization: The Third Xiangya Hospital of Central South University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021HP
Record Dates: First submitted 2021-10-16; First posted 2021-10-28 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Amoxicillin; Doxycycline; Furazolidone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group1: Vonoprazan Fumarate + amoxicillin + doxycycline (Experimental)
  Interventions: Drug: Group1 Vonoprazan Fumarate + amoxicillin + doxycycline
- Group2: Vonoprazan Fumarate + furazolidone + doxycycline (Experimental)
  Interventions: Drug: Group2 Vonoprazan Fumarate + furazolidone + doxycycline
- Group3: esomeprazole + colloidal bismuth tartrate + amoxicillin + doxycycline (Experimental)
  Interventions: Drug: Group3 esomeprazole + colloidal bismuth tartrate + amoxicillin + doxycycline
- Group4: esomeprazole + colloidal bismuth tartrate + furazolidone + doxycycline (Experimental)
  Interventions: Drug: Group4 esomeprazole + colloidal bismuth tartrate + furazolidone + doxycycline

INTERVENTIONS:
Drug: Group1 Vonoprazan Fumarate + amoxicillin + doxycycline — Vonoprazan Fumarate + amoxicillin + doxycycline
  Arms: Group1: Vonoprazan Fumarate + amoxicillin + doxycycline
Drug: Group2 Vonoprazan Fumarate + furazolidone + doxycycline — Vonoprazan Fumarate + furazolidone + doxycycline
  Arms: Group2: Vonoprazan Fumarate + furazolidone + doxycycline
Drug: Group3 esomeprazole + colloidal bismuth tartrate + amoxicillin + doxycycline — esomeprazole + colloidal bismuth tartrate + amoxicillin + doxycycline
  Arms: Group3: esomeprazole + colloidal bismuth tartrate + amoxicillin + doxycycline
Drug: Group4 esomeprazole + colloidal bismuth tartrate + furazolidone + doxycycline — esomeprazole + colloidal bismuth tartrate + furazolidone + doxycycline
  Arms: Group4: esomeprazole + colloidal bismuth tartrate + furazolidone + doxycycline

SUMMARY:
To compare the performance of four treatment regimens for radical treatment of Helicobacter pylori, evaluating the efficacy, safety, patient compliance, and socioeconomic evaluation of the four regimens. The four treatment regimens included (1) Vonoprazan Fumarate + amoxicillin + doxycycline, (2) Vonoprazan Fumarate + furazolidone + doxycycline, (3) esomeprazole + colloidal bismuth tartrate + amoxicillin + doxycycline, and (4) esomeprazole + colloidal bismuth tartrate + furazolidone + doxycycline.

DETAILED DESCRIPTION:
A single-center, prospective, open-label, parallel control design was conducted to enroll 100 patients with confirmed Helicobacter pylori infection. Patients were randomly divided into four groups, respectively accept four treatment regimens including (1) Vonoprazan Fumarate + amoxicillin + doxycycline, (2) Vonoprazan Fumarate + furazolidone + doxycycline, (3) esomeprazole + colloidal bismuth tartrate + amoxicillin + doxycycline, and (4) esomeprazole + colloidal bismuth tartrate + furazolidone + doxycycline. The effectiveness, safety and compliance of the four regimens were compared, and the cost-benefit analysis of the different regimens was conducted. The purpose of this study was to explore the most appropriate treatment plan for radical treatment of Helicobacter pylori .

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, ≤80 years
2. Urea breath test (UBT) was positive for Hp infection;
3. WIthout any anti-Hp treatment before
4. Endoscopy was performed within 1 month
5. Understanding the purpose and procedure of the study, voluntarily participating in the study and signing a written informed consent.

Exclusion Criteria:

1. Allergic to drugs used in this clinical study;
2. Using PPI, histamine H2 receptor antagonist, antibiotics, bismuth, probiotics or drugs with antibacterial effects within 4 weeks before treatment.
3. Using adrenal corticosteroids, non-steroidal anti-inflammatory drugs and anticoagulants
4. The disease or clinical condition that may interfere with the treatment evaluation of the study, such as liver disease, cardiovascular disease, lung disease, kidney disease, metabolic disease, psychiatric disease, or malignant tumor
5. Pregnant or lactating women
6. Participated in other clinical studies within 3 months prior to the registration of this clinical study
7. Suspected history of antibiotic abuse
8. Patients with craniocerebral injury, mental illness or epilepsy who cannot communicate with others or other diseases that may affect follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-17 (Actual); Primary Completion 2022-06-17 (Estimated); Study Completion 2022-10-17 (Estimated)

PRIMARY OUTCOMES:
Eradication rate of Hp at one time | 43 or 57 days after the initiation of eradication therapy
  The UBT test was performed to determine whether Hp was eradicated. No antibiotics, bismuth, or PPI were taken during this period. ITT analysis and PP analysis were used.

SECONDARY OUTCOMES:
Cost-benefit analysis | 43 or 57 days after the initiation of eradication therapy
  The drug cost of the two treatment options was calculated. According to the HP eradication rate, markov model was used to conduct cost-benefit analysis of the two methods, and determine which method was more cost-effective from an economic perspective.
Adverse events | 43 or 57 days after the initiation of eradication therapy
  Adverse drug events, significant laboratory outliers, and new diseases emerging during the study

CONTACTS AND LOCATIONS:
Locations (1):
- The third Xiangya Hospital of central south University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Z, Liu F, Ai F, Chen X, Liu R, Zhang C, Fang N, Fu T, Wang X, Tang A. The efficacy and mechanism of vonoprazan-containing triple therapy in the eradication of Helicobacter pylori. Front Pharmacol. 2023 May 5;14:1143969. doi: 10.3389/fphar.2023.1143969. eCollection 2023. PMID 37214450

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-05-23): https://cdn.clinicaltrials.gov/large-docs/46/NCT05097846/Prot_SAP_ICF_001.pdf